CLINICAL TRIAL: NCT00002333
Title: A Randomized, Double-Blind, Multicenter, Parallel Study of Ro 31-8959 (Saquinavir; HIV Proteinase Inhibitor) Alone, HIVID (Dideoxycytidine; Zalcitabine, ddC) Alone, and Both in Combination, as Treatment for Advanced HIV Infection (CD4 50-300 Cells/mm3) in Patients Discontinuing or Unable to Take Retrovir (Zidovudine; AZT) Therapy
Brief Title: A Study of Saquinavir and Zalcitabine, Used Alone and Together, in the Treatment of Advanced HIV Infection in Patients Who Stopped Taking or Who Cannot Take Zidovudine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 229A; NV 14256B; NV 14256A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-02

CONDITIONS: HIV Infections
Keywords: Zalcitabine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Saquinavir; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Saquinavir; Zalcitabine

INTERVENTIONS:
Drug: Saquinavir
Drug: Zalcitabine

SUMMARY:
To compare the safety, tolerance, and efficacy of saquinavir mesylate (Ro 31-8959) alone, zalcitabine (dideoxycytidine; ddC) alone, and both in combination, in patients discontinuing or unable to take zidovudine (AZT).

DETAILED DESCRIPTION:
Patients are randomized to one of three treatment regimens: ddC alone, Ro 31-8959 alone, and ddC plus Ro 31-8959. Treatment continues for at least 48 weeks. Patients are stratified by baseline CD4 count. (Per 09/26/94 amendment, a fourth arm, lower dose Ro 31-8959 plus ddC, was discontinued.)

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* G-CSF and erythropoietin.
* Prophylaxis or chronic suppression/maintenance therapy with dapsone, aerosolized pentamidine, isoniazid, rifampin, fluoroquinolones, pyrazinamide, ethambutol, fluconazole, itraconazole, acyclovir, clotrimazole, nystatin, trimethoprim/sulfamethoxazole, pyrimethamine, folic acid, sulfadiazine, clindamycin, and fansidar.

Concurrent Treatment:

Allowed:

* Limited localized radiation therapy to the skin.

Patients must have:

* Documented HIV infection.
* CD4 count 50 - 300 cells/mm3.
* Received prior AZT that has been discontinued at least 28 days prior to study entry.
* No active opportunistic infection requiring immediate treatment.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Signs or symptoms of peripheral neuropathy.
* Malabsorption or inadequate oral intake (defined as unable to eat one or more meals daily because of chronic nausea, emesis, or abdominal/oral-esophageal discomfort.
* Malignancy, visceral Kaposi's sarcoma, or lymphoma requiring systemic chemotherapy and/or radiotherapy within the next 48 weeks.
* Any grade 3 or worse laboratory or clinical abnormality.
* Inability to comply with protocol requirements.

Concurrent Medication:

Excluded:

* Other antiretroviral drugs.
* Experimental drugs.
* Nephrotoxic or hepatotoxic drugs.
* Drugs likely to cause peripheral neuropathy.
* Antineoplastic agents.
* Biologic response modifiers.

Concurrent Treatment:

Excluded:

* Radiation therapy other than limited localized therapy to skin.

Patients with the following prior conditions are excluded:

* History of non-Hodgkin's lymphoma.
* Unexplained fever >= 38.5 C (101.5 F) persisting for 14 days or longer within the 28 days prior to study entry.
* Unexplained, chronic diarrhea (defined as 3 or more loose stools daily) persisting for 14 days or longer within the 28 days prior to study entry.
* History of grade 2 or worse peripheral neuropathy.

Prior Medication:

Excluded:

* Prior HIV proteinase inhibitor.
* Prior antiretroviral therapy other than AZT.
* Acute therapy for opportunistic infection within 14 days prior to study entry.

Prior Treatment:

Excluded:

* More than 3 units of blood in any 21-day period within 3 months prior to study entry.

Required:

* Prior AZT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900

CONTACTS AND LOCATIONS:
Locations (47):
- United States (41):
  - Kaiser Foundation Hosp, Harbor City, California
  - UCSD, La Jolla, California
  - UCLA School of Medicine, Los Angeles, California
  - CARE Ctr / UCLA Med Ctr, Los Angeles, California
  - UCD, Sacramento, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Davies Med Ctr / c/o HIV Institute, San Francisco, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - San Francisco Veterans Administration Med Ctr, San Francisco, California
  - Pacific Oaks Med Group / Rsch & Scientific Investigation, Sherman Oaks, California
  - Sunnyvale Med Clinic, Sunnyvale, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Veterans Administration Med Ctr, Washington D.C., District of Columbia
  - Miami Veterans Administration Med Ctr, Miami, Florida
  - Univ of Miami Dept of Medicine, Miami, Florida
  - Stratogen of South Florida, Miami Beach, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - West Paces Clinical Research Incoporated, Atlanta, Georgia
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Tulane Univ Med School, New Orleans, Louisiana
  - New England Med Ctr, Boston, Massachusetts
  - Massachusetts Gen Hosp / Harvard Med School, Boston, Massachusetts
  - New England Deaconess Hosp, Boston, Massachusetts
  - Harper Hosp, Detroit, Michigan
  - Washington Univ School of Medicine, St Louis, Missouri
  - UMDNJ - New Jersey Med School / Cooper Hosp, Camden, New Jersey
  - UMDNJ - New Jersy Med School, Newark, New Jersey
  - Albany Med College, Albany, New York
  - Beth Israel Med Ctr, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Harkness Pavilion, New York, New York
  - Ohio State Univ Hosp, Columbus, Ohio
  - Oregon Health Sciences Univ, Portland, Oregon
  - Thomas Jefferson Med College, Philadelphia, Pennsylvania
  - Graduate Hosp / Tuttleman Cancer Ctr, Philadelphia, Pennsylvania
  - Univ of Tennessee, Memphis, Tennessee
  - Oaklawn Physicians Group, Dallas, Texas
  - Univ TX Galveston Med Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Univ of Washington / Harborview Med Ctr, Seattle, Washington
- Canada (5):
  - Southern Alberta HIV Clinic, Calgary, Alberta
  - McMaster Univ Med Ctr, Hamilton, Ontario
  - Sunnybrook Health Science Ctr, Toronto, Ontario
  - Clinique Medicale L'Actuele, Montreal, Quebec
  - Montreal Gen Hosp, Montreal, Quebec
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Revicki D, Swartz C. Quality of life outcomes of saquinavir, zalcitabine and combination saquinavir-zalcitabine therapy for advanced HIV-infection. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:113 (abstract no 266)